CLINICAL TRIAL: NCT04635176
Title: Infiltration Between the Popliteal Artery and the Capsule of the Knee (iPACK) With Local Infiltration of Analgesia (LIA) and Adductor Canal Block (ACB) Improves Postoperative Pain in Total Knee Arthroplasty: A Randomized Controlled Trial
Brief Title: Comparing Local Anesthesia With and Without iPACK Block
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Alberta Health services (Other); Alberta Hip and Knee Clinic (Other)
Responsible Party: Principal Investigator, Rajrishi Sharma, Assistant Clinical Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: "REB20-1633"
Record Dates: First submitted 2020-10-23; First posted 2020-11-18 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Osteo Arthritis Knee; Analgesia; Pain, Postoperative
MeSH Terms: conditions — Agnosia; Pain, Postoperative | interventions — Bupivacaine; Epinephrine; Anesthesia, Local; Saline Solution

STUDY DESIGN:
Intervention Model Description: Group A will receive perioperative ACB, LIA, and sham IPACK block. Group B will receive perioperative ACB, LIA, and real IPACK block.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study personnel, including research team, anesthesiologists, surgeons, physiotherapists, recovery room and ward nurses, as well as patients will be blinded to the group allocation. Anesthesia assistants not involved in study data collection or patient care will prepare the sham or real local anesthetic injectate solution for iPACK block. Syringes will be prepared immediately after randomization and before block placement and provided to the blinded anesthesiologist.
  The statistician who run randomization would only know study IDs and stay blinded to patients' treatment arms.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sham iPACK block (Placebo Comparator): This groups will receive the adductor canal block with the local anesthetic (15 mL of 0.25% bupivacaine + 2.5 mcg/mL epinephrine + 50 mcg/mL preservative-free dexamethasone) and local infiltration of analgesia+ sham iPACK block with 20 mL of normal saline.
  Interventions: Drug: Sham iPACK block with 20ml normal saline
- Real IPACK block. (Active Comparator): This groups will receive the adductor canal block with the local anesthetic (15 mL of 0.25% bupivacaine + 2.5 mcg/mL epinephrine + 50 mcg/mL preservative-free dexamethasone) and local infiltration of analgesia + real iPACK block with 20 mL of 0.25% bupivacaine, 2.5mcg/mL epinephrine, and 50mcg/mL preservative-free dexamethasone
  Interventions: Drug: Real iPACK block (20 mL of 0.25% bupivacaine, 2.5mcg/mL epinephrine, and 50mcg/mL preservative-free dexamethasone)

INTERVENTIONS:
Drug: Real iPACK block (20 mL of 0.25% bupivacaine, 2.5mcg/mL epinephrine, and 50mcg/mL preservative-free dexamethasone) — real iPACK block with 20 mL of 0.25% bupivacaine, 2.5mcg/mL epinephrine, and 50mcg/mL preservative-free dexamethasone
  Other Names: real iPACK block with local anesthesia
  Arms: Real IPACK block.
Drug: Sham iPACK block with 20ml normal saline — Sham iPACK block with 20 ml Normal saline
  Other Names: sham iPACK block with Normal saline
  Arms: Sham iPACK block

SUMMARY:
Total knee arthroplasty is an effective surgical intervention for patients with chronic osteoarthritis commonly performed worldwide. Postoperative pain management has been a key focus in patient care for this procedure. Poorly controlled pain following total knee arthroplasty is associated with decreased ambulation, increased length of hospital stay, increased complications (particularly related to significant opioid use), and overall suboptimal patient recovery. Appropriate postoperative pain management utilizing motor sparing peripheral nerve blocks and periarticular injections has been shown to provide faster, more optimized patient recovery and reduced hospital length of stay in patients undergoing total knee arthroplasty.

Adductor canal block (ACB) is a well-studied peripheral nerve block performed for analgesia following total knee arthroplasty. ACB is an effective component of multimodal analgesia providing improved pain control to the peripatellar and intra-articular aspect of the knee joint while largely preserving the strength of the quadriceps muscles1. In addition, perioperative local infiltration analgesia (LIA) performed by the orthopaedic surgical team is a common practice that has been shown to improve short-term postoperative pain relief and reduce total systemic opioid consumption during hospital stay2 for total knee arthroplasty.

The Infiltration between the Popliteal Artery and Capsule of the Knee (iPACK) block is a newly described regional anesthesia technique for postoperative analgesia in total knee arthroplasty, performed under ultrasound guidance. It targets the articular branches of the tibial, common peroneal, and obturator nerves in the popliteal region, and aims to provide analgesia to the posterior aspect of the knee joint without compromising lower extremity motor function following total knee arthroplasty.

This study aims to determine whether the IPACK block provides additional analgesia (in combination with ACB + LIA) for total knee arthroplasty surgeries. The study will examine how much additional analgesia IPACK provides in the context of an already-optimized regional anesthesia pathway for total knee arthroplasty, which uses ACB + LIA, both modalities that have reasonable existing evidence.

DETAILED DESCRIPTION:
Currently, limited studies exist in the literature regarding the use of iPACK for analgesia in total knee arthroplasty. Specific studies on the addition of iPACK to ACB or LIA demonstrate clinically significant reductions in pain scores for patients undergoing total knee arthroplasty. However, no studies currently examine the use of iPACK in the setting of patients receiving both ACB and LIA, as a fully optimized regional anesthesia "bundle" for postoperative analgesia in total knee arthroplasty. As such, this study aims to determine whether the addition of the iPACK block, in combination with ACB and LIA, will improve analgesia compared to what is provided by ACB and LIA alone.

Rationale for study:

The IPACK block, based on limited existing literature, seems to provide superior analgesia with minimal complications following total knee arthroplasty.

This study aims to determine whether the IPACK block provides additional analgesia (in combination with ACB + LIA) for total knee arthroplasty surgeries. The study will examine how much additional analgesia IPACK provides in the context of an already-optimized regional anesthesia pathway for total knee arthroplasty, which uses ACB + LIA, both modalities that have reasonable existing evidence.

Determining the effectiveness of IPACK in addition to the already validated multimodal analgesia including ACB and LIA for improving postoperative pain may further improve clinical outcomes in patients undergoing total knee arthroplasty. This may reduce postoperative opioid requirements and its side effects, increase patient satisfaction, and decrease morbidity and mortality associated with a prolonged hospital stay.

The demand for total knee arthroplasty is predicted to increase in the upcoming years owing to an aging population and increased prevalence of osteoarthritis worldwide. The growing number generates multiple issues to the healthcare system, mainly the additional pressure to decrease the already unsustainable high healthcare costs. The role of iPACK as an additional component of pain management may be the key to providing a safe and cost-effective healthcare service to patients undergoing total knee arthroplasty.

Study Question Does the addition of the iPACK block, in combination with ACB and LIA, improve postoperative analgesia and clinical outcomes compared to ACB and LIA alone in patients undergoing total knee arthroplasty?

Hypothesis:

Investigators hypothesize that the addition of this newly described, motor-sparing iPACK block will significantly improve analgesia and clinical outcomes in patients undergoing total knee arthroplasty.

Study Design :

To determine the effectiveness of the iPACK block as a component of multimodal analgesia for patients undergoing total knee arthroplasty, this study will be a prospective double blinded randomized controlled trial where the patients will be randomized to 2 groups:

Group A will receive perioperative ACB, LIA, and sham IPACK block. Group B will receive perioperative ACB, LIA, and real IPACK block.

In addition, all patients will receive a standard spinal anesthetic as per our institutional protocol, along with procedural IV sedation at the discretion of the attending anesthesiologist. Local infiltration analgesia will be administered by the orthopaedic surgeon as per standard practice. ACB and iPACK block will be performed by the anesthesiologist immediately preoperatively under ultrasound guidance as follows:

All patients in the study will receive ACB, performed by an experienced anesthesiologist, as conventionally described, using full aseptic technique, in-plane ultrasound guidance, identification of the superficial femoral artery, sartorius muscle and adductor canal. Local anesthetic (0.25% bupivacaine + 2.5mcg/mL epinephrine + 50mcg/mL preservative-free dexamethasone x 15mL) will be infiltrated with real-time ultrasound visualization, needle approach lateral to medial, with incremental injection, intermittent aspiration, and confirmation of adequate local anesthetic spread.

Patients in group A will receive a sham iPACK block while those in group B will receive a real iPACK block. Both sham and real iPACK blocks will be performed by an experienced anesthesiologist, blinded to the intervention. Real and sham iPACK blocks will be performed as conventionally described with ultrasound guidance (initial approach 1 finger breadth above the patella, if this approach fails, subsequent attempt at level of femoral condyles/bicondylar approach). All sham and real iPACK blocks will be done with full aseptic technique, in-plane ultrasound guidance, identification of popliteal artery/vessels, femur, and sciatic nerve. Normal saline x 20mL (Group A), or local anesthetic x 20mL (Group B - 0.25% bupivacaine + 2.5mcg/mL epinephrine + 50mcg/mL preservative-free dexamethasone), will be infiltrated with real-time ultrasound visualization, needle approach medial to lateral, with incremental injection, intermittent aspiration, and confirmation of adequate local anesthetic spread.

The study personnel, including research team, anesthesiologists, surgeons, physiotherapists, recovery room and ward nurses, as well as patients will be blinded to the group allocation. Anesthesia assistants not involved in study data collection or patient care will prepare the sham or real local anesthetic injectate solution for iPACK block. Syringes will be prepared immediately after randomization and before block placement and provided to the blinded anesthesiologist. Pain scores and opioid consumption, length of stay, and other data will be collected and assessed in person by a member of the research team or patient care team who is blinded to study interventions.

Study procedure:

Participating orthopaedic surgeons will identify eligible patients and introduce them to the study and research team at Alberta Hip and Knee Clinic (AHKC). Research staff will follow recruitment procedure and seek informed consent from patients at AHKC. Participation in this study will remain completely voluntary without any pressure from investigators. Patients' questions will be answered at recruitment session. Upon recruitment, patients will be asked to complete Western Ontario and McMaster Universities Arthritis Index (WOMAC) and Knee Society Scoring (KSS).

Study participants will be assigned study identification and get randomized in to two treatment arms.

The statistician who run randomization would only know study identifications and stay blinded to patients' treatment arms. Hospital data will be used to know Length of Stay (LOS) and opioid consumption at hospital. A physiotherapist will perform Timed Up and Go test and Range of Motion (ROM) Pre and post-operatively at Peter Lougheed Hospital. Pain score will be recorded using Visual analogue scale 4 hours postoperatively and at discharge. Emergency room visit or 30-day readmission will be accessed through Alberta Bone and Joint Health Institute (ABJHI) data repository. "Unanticipated complications of iPACK block" and "technical difficulties with performing the iPACK block" will be recorded by the study anesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective unilateral TKA
* Planned for regional anesthesia for the procedure
* Age >=18

Exclusion criteria:

* Contraindications to regional anesthesia or peripheral nerve blocks
* Allergy to local anesthetics or any of the study medications
* Severe hepatic or renal insufficiency
* Chronic opioid consumption
* Patient with difficulty comprehending visual analogue scale pain scores
* Pre-existing lower extremity neurologic abnormalities
* Patients classified as American Society of Anesthesiologists score 3 or 4
* Language/communication barrier

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2022-10-30 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Comparing pain scores using the visual analogue scale between 2 groups | 4 hours after surgery
  Visual analogue scale is a tool to measure intensity of pain in human. It is numeric (0-100);A higher score indicates greater pain intensity.
Comparing pain scores using the visual analogue scale between 2 groups | 24 hours after surgery
  Visual analogue scale is a tool to measure intensity of pain in human. It is numeric (0-100);A higher score indicates greater pain intensity.
Comparing total opioid consumption between 2 groups | During 24 hours after surgery
  Opioid consumption will be compared between two groups by measuring how many milligrams opioids patients consume in each group, the total dose of opioids consumed by patients will be converted to oral morphine dose equivalents in milligrams, and this mg value will be compared between the groups. The opioid can refer to morphine or oxycodone or hydromorphone or codeine any kind of opioid-type medication. There is a standard conversion of any other opioid potency to "morphine equivalents" (eg: hydromorphone is 5x more potent than morphine).
Comparing total length of hospital stay | 20-48 hours after surgery
  Comparing total length of hospital stay
Timed Up and Go test results | pre-intervention
  Timed Up and Go test results
Timed Up and Go test results | Up to 24 hours after surgery
  Timed Up and Go test results
Comparing knee Range of Motion (ROM) | pre-intervention
  Comparing knee Range of Motion (ROM)
Comparing knee Range of Motion (ROM) | Up to 24 hours after surgery
  Comparing knee Range of Motion (ROM)
Comparing patient satisfaction using Western Ontario and McMaster Universities Arthritis Index (WOMAC) | Up to 24 hours after surgery
  The WOMAC is a patient reported outcome questionnaire, consisting 24 items divided into three subscales: 1) Pain (5 items), 2) Stiffness (2 items) and 3) Physical Function (17 items). A total WOMAC score is created by summing the items for all three subscales. Higher scores on the WOMAC indicate worse pain, stiffness, and functional limitations. Previous assessment has supported the internal consistency of the WOMAC subscale.
Comparing patient satisfaction using Knee Society Scoring (KSS) | Up to 24 hours after surgery
  The Knee Society Scoring system is both physician and patient-derived. It includes versions to be administered pre-operatively and post-operatively. It has an initial assessment of demographic details, including an expanded Charnley Functional classification. The objective knee score, completed by surgeon, includes a Visual Analogue Scale score of pain walking on level ground and on stairs or inclines, as well as an assessment of alignment, ligament stability, and Range Of Motion. The KSS System is a validated instrument based on surgeon and patient generated data, adapted to the diverse lifestyles and activities. The greater score associated with higher satisfaction.

SECONDARY OUTCOMES:
Number pf participants returning to emergency room in the hospital | Within 30 days after surgery
  Number pf participants returning to emergency room in the hospital
Incidence of the unanticipated motor block from iPACK intervention by a questionnaire filled out by the attending anesthesiologist | Up to 24 hours after surgery
  Incidence of the unanticipated motor block from iPACK intervention by a questionnaire filled out by the attending anesthesiologist
Incidence of other unanticipated complications of iPACK intervention by a questionnaire filled out by the attending anesthesiologist | Up to 24 hours after surgery
  Incidence of other unanticipated complications of iPACK intervention by a questionnaire filled out by the attending anesthesiologist
Incidence of technical difficulties experienced by a questionnaire filled out by the attending anesthesiologist on the day of surgery | 24 hours after surgery
  Incidence of technical difficulties experienced by a questionnaire filled out by the attending anesthesiologist on the day of surgery
Comparing duration (in minutes) of tourniquet use during surgery between two groups | During surgery time
  Tourniquets are tight bands used to completely stop the blood flow to a wound. Duration of its use will be noted at operation room in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Rajrishi Sharma, MD, Principal Investigator — University of Calgary
Locations (1):
- University of Calgary/AB Hip and Knee Clinic, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No